CLINICAL TRIAL: NCT06047665
Title: Tracheostomy Decannulation Outcomes: A Longitudinal Observational Study
Brief Title: Outcomes After Tracheal Cannula Removal
Acronym: Dekan
Status: Recruiting | Type: Observational
Sponsor: Katharina Winiker (Other)
Collaborators: Swiss Paraplegic Research, Nottwil (Network)
Responsible Party: Sponsor-Investigator, Katharina Winiker, Principal Investigator, Swiss University of Speech and Language Sciences
Organization: Swiss University of Speech and Language Sciences (Other)
Other Study IDs: 2022-08
Record Dates: First submitted 2023-08-30; First posted 2023-09-21 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Tracheostomy
Keywords: Tracheostomy; Decannulation; Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This longitudinal observational study involves an integrated knowledge translation (IKT) approach involving key stakeholders in the project team to evaluate the tracheostomy management in patients hospitalized in the Swiss Paraplegic Centre Nottwil (SPC).

DETAILED DESCRIPTION:
Primary objective

- to evaluate the rate of physical complications (that require treatment, intubation, recannulation or lead to death) in patients hospitalized in the SPC over three months following the removal of the tracheal cannula (decannulation).

Secondary objectives

* to describe types of complications short-term (up to 4 days) and long-term (up to three months) post-decannulation
* to assess predictors for short- and long-term complications post-decannulation
* to explore patients' perspectives on decannulation outcomes
* to evaluate individual trajectories of the clinical decannulation protocol

ELIGIBILITY:
Inclusion Criteria:

* at the time of recruitment, tracheotomized adult in-patients (≥ 18 years) of the SPC with any medical diagnosis
* decannulated in the Swiss Paraplegic Center Nottwil within the project's data collection period
* German, French, Italian or English as communication language
* study consent

Exclusion Criteria:

* patients for whom no decannulation is sought (e.g., due to degenerative illness)
* patients for whom decannulation is planned in a clinic other than the SPC (e.g., patients hospitalized in the SPC for weaning only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Tracheotomized patients hospitalized in the Swiss Paraplegic Centre Nottwil.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-08-25 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
rate of physical complications post-decannulation | for 3 months post-decannulation (assessment time points: 4 days, 1 month, and 3 months post-decannulation)
rate of reintubation post-decannulation | for 3 months post-decannulation (assessment time points: 4 days, 1 month, and 3 months post-decannulation)
rate of recannulation post-decannulation | for 3 months post-decannulation (assessment time points: 4 days, 1 month, and 3 months post-decannulation)
rate of death post-decannulation | for 3 months post-decannulation (assessment time points: 4 days, 1 month, and 3 months post-decannulation)

SECONDARY OUTCOMES:
types of decannulation-related physical complications short- and long-term | for 3 months post-decannulation (assessment time points: 4 days, 1 month, and 3 months post-decannulation)
  including excessive secretion, altered respiratory frequency, respiratory insufficiency, respiratory infections, newly occuring neurological symptoms, sleep apnea, intratracheal complications, complications with tracheostoma
candidate prognostic factors for physical complications post-decannulation | 1 week pre-decannulation, (4 days for one select parameter), 1 month, and 3 months post-decannulation
  individual demographic and clinical patient characteristics
patients' perspectives on decannulation outcomes | Questionnaire: 4 days, 1 month, and 3 months post-decannulation; Human Flourishing Measure: 1 week pre-decannulation and 3 months post-decannulation
  A questionnaire will be used to assess advantages and disadvantages of the decannulation (8 questions, per question 3 - 6 pre-formulated answers to choose from). Additional, the Harvard Human Flourishing Measure (12 questions, rating from 0 to 10 per question, sum score to calculate the 'flourish measure') will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Katharina Winiker, PhD, Principal Investigator — Swiss University of Speech and Language Sciences; Gabi Müller Verbiest, PhD, Study Chair — Swiss Paraplegic Center Nottwil
Locations (1):
- Swiss Paraplegic Center Nottwil, Nottwil, Canton of Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Winiker K, Stierli S, Brinkhof MWG, Hamzic S, Schwegler H, Mueller G. Outcomes of Tracheostomy Decannulation: Study Protocol for a Longitudinal Observational Study. Int J Lang Commun Disord. 2026 Jan-Feb;61(1):e70165. doi: 10.1111/1460-6984.70165. PMID 41355759